CLINICAL TRIAL: NCT05540132
Title: Slow-digestible Carbohydrates Consumed Prior to Exercise Improve Performance and Decrease Risk of Delayed Hypoglycemia in Adolescents with Type 1 Diabetes
Brief Title: Slow Digestible Carbohydrates and Exercise in Adolescents with Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Lucy D Mastrandrea, Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SS_T1D_2022
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: adolescent; exercise; cgm
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Within subject, randomized cross-over study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast Acting Carbohydrate (Active Comparator): Prior to exercise performance test, subject will be randomized to consume 22 grams of fast-acting carbohydrate (maltodextrin) or slow-acting cornstarch based supplement
  Interventions: Dietary Supplement: maltodextrin
- Slow-acting cornstarch supplement (Active Comparator): Prior to exercise performance test, subject will be randomized to consume 22 grams of slow-acting cornstarch based supplement or fast-acting carbohydrate (maltodextrin)
  Interventions: Dietary Supplement: super starch

INTERVENTIONS:
Dietary Supplement: maltodextrin — Pre-exercise carbohydrate, fast-acting
  Arms: Fast Acting Carbohydrate
Dietary Supplement: super starch — Pre-exercise carbohydrate, slow-acting
  Arms: Slow-acting cornstarch supplement

SUMMARY:
In this within-subject cross-over study, the investigators hypothesize that corn-starch based supplements taken prior to exercise will decrease the risk of delayed hypoglycemia in adolescents with T1D, improve performance during exercise, and decrease glycemic variability during exercise.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D), one of the most common chronic diseases in adolescents, is caused by the destruction of insulin producing beta cells which are located in the pancreas. There are many factors that impact diabetes control which are insulin administration, intake of food and exercise. When an individual exercises, weight is better managed which allows for a better cardiovascular system. Exercising also improves insulin sensitivity which can increased the risk for delayed hypoglycemia (low blood sugar). Many individuals with T1D do not participate (or under-participate) in exercise due to the fear of hypoglycemia. This study will recruit adolescents with Type 1 diabetes to undergo a maximal exercise test to determine their VO2max. Study participants then will complete 2 exercise performance tests prior to which the participant will be randomized to consume 22 grams of either fast acting carbohydrates or long-acting cornstarch based supplements. Subjects will be asked to bike for 45 minutes (at 50% of VO2max) and then complete a 3.75 mile bike ride as quickly as possible. The investigators will document the time to completion of the bike ride as well as monitor glucose levels via continuous glucose monitoring for 12 hours after completion of the exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - <18 year old male and female subjects with Type 1 diabetes for > 1 year
* HbA1c <10.5%
* Body Mass Index >10th % and <95th%
* Not being treated with sensor-augmented pump therapy
* Ability to participate in exercise activity - biking
* Willing to wear a continuous glucose monitor (CGM) sensor

Exclusion Criteria:

* Severe hypoglycemia (requiring glucagon or external assistance) in last 6 months
* Admission for diabetic ketoacidosis in last 3 months
* History of chronic lung disease, congenital heart disease or chronic asthma
* Food (including corn)/dye allergies
* Other chronic medical conditions except for well-controlled thyroid disease

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — All genders are eligible, patients self-identification of gender will be recorded
Enrollment: 20 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of hypoglycemic events 12 hours after completion of exercise challenge | 12 hours after exercise challenge
  Review of continuous glucose monitoring data
Glycemic variability during exercise challenge | During exercise challenge
  Review of continuous glucose monitoring data
Time to completion of distance bike challenge | During exercise challenge
  Number of minutes to complete 3.75 mile bike ride

SECONDARY OUTCOMES:
Percent time spent in hypoglycemia following exercise challenge | 12 hours after exercise challenge
  Review of continuous glucose monitoring data
Percent time above range, in range, and below range following exercise challenge | 12 hours after exercise challenge
  Review of continuous glucose monitoring data
Glycemic variability in the 12 hours following the exercise test | 12 hours after exercise challenge
  Review of continuous glucose monitoring data

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Mastrandrea, MD, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- UB MD Pediatrics Division of Pediatric Endocrinology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Consent informs subjects as follows:
  If identifiers are removed from your identifiable information, that information could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent. Any future use of the banked data for research outside the scope of this current protocol will be submitted as separate studies to the Institutional Review Board for review and approval, prior to conducting the research
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available June, 2024 and will be available for 2 years
Access Criteria: Contact with Principal Investigator